CLINICAL TRIAL: NCT04267809
Title: Modulating Endoplasmic Reticulum Stress as a Prophylactic Approach Against Symptomatic Viral Infection
Brief Title: Modulate Cellular Stress in the Immune Cells to Reduce Rate of Symptomatic Viral Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Met-YF-001
Record Dates: First submitted 2020-02-05; First posted 2020-02-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Endoplasmic Reticulum Stress; Viral Infection; Yellow Fever
Keywords: Metformin; Endoplasmic Reticulum Stress; YF17D infection; Symptomatic; Metabolic; Immunometabolism
MeSH Terms: conditions — Virus Diseases; Yellow Fever | interventions — Metformin; Calcium; Vitamin D

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized into one of two groups in the same ratio (1:1). As this is an open-label study, random block sizes will be used to avoid selection bias yet ensure balance over time. Randomization will be performed via a web-based randomization system: http://www.randomization.com by an independent person who has no direct contact with the subjects. Randomization opaque envelopes will be prepared by an independent team in accordance to the Master Randomization List generated. The randomization envelopes are to be opened sequentially for each enrollment by the study team and will determine the subject's allocation to one of the two groups.
Who Masked: Participant, Investigator
Masking Description: This is a randomized, double-blind, placebo-controlled clinical trial of metformin in 44 healthy adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): 22 subjects will receive Metformin 1000mg twice daily for 7 consecutive days (Days 1-7). On Day 4, subjects will be administered one dose of YF17D before metformin dosing.
  Interventions: Drug: Metformin Hydrochloride
- Placebo group (Placebo Comparator): 22 subjects will receive placebo twice daily for 7 consecutive days (Days 1-7). On Day 4, subjects will be administered one dose of YF17D before placebo dosing.
  Interventions: Drug: Calcium and Vitamin D

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin 500mg tablets are registered and licensed in Singapore. For the study, we will be sourcing the Metformin tablets from Singapore General Hospital Formulary.
  Other Names: Metformin
  Arms: Metformin group
Drug: Calcium and Vitamin D — Calcium and Vitamin D tablets are registered and licensed in Singapore. For the study, we will be sourcing the Calcium and Vitamin D tablets from Singapore General Hospital Formulary.
  Arms: Placebo group

SUMMARY:
To determine the efficacy of metformin in reducing the rate of symptomatic YF17D infection, and to elucidate the effects of metformin on YF17D viremia and the downstream adaptive immune response, we hereby propose a randomised, double-blind, placebo-controlled clinical trial that is coupled with a system biology approach. We plan to recruit 44 healthy volunteers aged 21-40 years, with a Body Mass Index of 20-25 kg/m2, have no known drug allergies and are not currently receiving regular immune-modulating therapy such as metformin, NSAIDs, paracetamol, corticosteroids or statins. The age range that we propose will ensure that our volunteers are likely to be healthy and not be on long-term medication for other concurrent medical conditions. This would abrogate the confounding effect of YF17D infection enhancement by cross reactive antibodies that we have previously shown.

Informed written consent will be obtained before any physical examination is performed. All consented subjects will undergo screening which includes a full physical examination, vital signs measurement, clinical laboratory tests and urine pregnancy test (for female subjects of child-bearing potential) Eligible subjects will be randomized 1:1 to either metformin 1000mg or placebo twice daily for 7 consecutive days (Days 1-7). On Day 4, subjects will be administered one dose of YF17D before study drug dosing.

Aim 1 tests the hypothesis that prophylactic metformin reduces ER stress and thus attenuates the post-infection pro-inflammatory response for reduced rate of symptomatic outcome. The primary objective for Aim 1 is to determine the efficacy of metformin in reducing the rate of symptomatic YF17D infection using a randomized placebo-controlled clinical trial.

Aim 2 explores the effectiveness of metformin, either through its action on ER stress or other pathways that differentially regulate the expression of pro- and anti-viral host factors, in inhibiting live attenuated vaccine infection and downstream adaptive immune responses. The primary objective for Aim 2 is to elucidate the effects of metformin on YF17D viremia and the downstream adaptive immune response.

DETAILED DESCRIPTION:
Criteria for Recruitment and Recruitment Process: Subjects will be recruited from SingHealth Investigational Medicine Unit (IMU) healthy volunteer database and recruitment posters. Subjects will be given a copy of the Participant Information and Informed Consent Form to read upon their arrival. A briefing session on the study will be conducted by the Investigator. Thereafter, subjects will be ushered into a private room where informed consent is obtained and where questions about the study can be asked freely. Subjects will not be rushed into making a decision to participate in the study. They will be encouraged to speak to their family members about participation in the study; and allowed to defer their decision (without any prejudice) to participate till after discussion with their family members.

Screening Visits and Procedures: Subjects will be recruited via the SingHealth Investigational Medicine Unit (IMU). Informed written consent will be obtained before any study related procedure or assessment is performed. All subjects' eligibility for recruitment into the study must be assessed during screening visit. Subjects must satisfy all inclusion and exclusion criteria outlined in Section 3.3 and Section 3.4 respectively to be eligible for enrolment into the study. Eligibility criteria must be confirmed before dosing. All clinical laboratory tests scheduled for screening will be collected to establish pre-dose baseline. Other procedures that must be completed before the study begins include a full physical examination and urinary pregnancy test (for female subjects of child-bearing potential).

Study Visits and Procedures: All eligible subjects will proceed to Day 1, where they will be randomized 1:1 to either metformin 1000mg or placebo twice daily for 7 consecutive days (Days 1-7). On Day 4, subjects will be administered one dose of YF17D before study drug dosing. Subjects will report to the SingHealth IMU on Day 1 (pre-study drug), Day 4 (pre-YF17D), Days 5, 7, 11, 14, 18 (only for participants who consent to scRNA-seq and T-cell studies) and Day 32 for research blood sampling. The schedule for blood draws will be identical for all study groups. All research blood samples will be stored at -80oC until recruitment is completed before analysis. Subject recruitment and blood collection will be conducted as an outpatient study in the SingHealth Investigational Medicine Unit (IMU), a dedicated early phase clinical trial facility. From our prior experience, we anticipate we will not have difficulty recruiting the required number of participants into our study necessary to meet our target sample size.

Post Study Follow up and Procedures: There is no requirement for post-study follow-up or procedures.

Safety Monitoring Plan: The study may be evaluated by government inspectors/regulatory authorities who must be allowed access to e-CRFs, source documents, and other study files. The inspectors will review CRFs and compare them with source documents to verify accurate and complete collection of data and confirm that the study is being conducted according to the protocol, ICH-Good Clinical Practices (ICH-GCP) and all applicable regulations.

Known common adverse events of metformin include diarrhoea, nausea, stomach pain, heartburn and bloatedness. Rare AEs include lactic acidosis and hypoglycaemia. Limiting the duration of metformin dosing to 10 days would further reduce the risk of these serious AEs. Subjects will be trained to look out for early symptoms associated with these AEs and to report to IMU immediately should they experience any of these symptoms. Details of AE event terminology, date and time of event start and end, severity, using the CTCAE or treatment given, impact on work and to the continuation of the study, and final outcome of the event will be recorded on the case report until resolution of the event.

During the study, the investigator will recruit the subjects, as well as perform full history taking and physical examination at both scheduled and unscheduled visits. The investigator will also review the subject's diaries for any potential side effects and manage the AEs based on best clinical practice should they arise. Compliance to study protocol will be checked by taking a medication history, and pill count and inspection of diary as well as measurement of metformin drug level at specific time points.

Data Quality Assurance: The PI and Co-Is will review the study periodically for data and safety monitoring. Internal quality checks will be performed by two CRCs who are study team members. The data entered by one CRC will be checked by another using the source documents. The study may also be picked for monitoring by SingHealth Office of Research Integrity and Compliance (ORIC) or evaluated by government inspectors/regulatory authorities who must be allowed access to e-CRFs, source documents, and other study files. The monitors/inspectors may review CRFs and compare them with source documents to verify accurate and complete collection of data and confirm that the study is being conducted according to the protocol, ICH-Good Clinical Practices (ICH-GCP) and all applicable regulations.

Data Entry and Storage: All participant's data will be de-identified upon recruitment. Hardcopy research data collection forms such as CRFs, logs and diaries will be kept in the Investigator's Site File and stored in SingHealth IMU under lock and key, accessible only to delegated study team members. Direct data capture of demographic and clinical data will be captured on source documents. Identifiers will be kept in a separate file in another office and every effort will be made to protect the privacy of the participants. The data to be analysed will contain only de-identified data. An electronic data capture system will be used. All electronic data will be password protected and can only be accessed by study team members. Specimens, test results or pathogen data will be stored at Duke-NUS EID laboratory in a stand-alone PC whereby access is password protected.

Determination of Sample Size: A sample size of 20 per arm will give 80% power to detect a reduction in systemic symptoms from 50% to 10% (risk difference = 0.4 reduction ratio = 0.8) in participants who receive placebo versus who are pre-treated with metformin versus placebo group at a 2-sided 5% type I error rate (PASS 13 Software). Factoring in a potential dropout rate of 10%, the total sample size is 44 in total (22 per arm). From our previous experience with subject recruitment in the YF vaccine trial, there were no dropouts during the 1-month follow-up period. Therefore, we are confident that we can recruit the required number of subjects within the trial period.

Statistical analysis: Fisher's exact test will be used to assess difference in systemic symptom rate between placebo and metformin pre-treatment arm. Confidence intervals (CI) for AE rates will be estimated using the exact method. CI for risk difference will be estimated using the Newcombe's score method.

Diagnostic plots will be used to determine the choice of using the raw data or log-transformed data in parametric analyses or non-parametric analyses. Differences in anti-YF neutralizing antibody titer at day 28, viremia and SBREP-1 expression will be compared between placebo and metformin groups. Relationship between systemic symptoms, molecular correlates of immunogenicity, viremia, antibody titer and metformin will be explored with regression methods. Differences in background characteristics between subjects who do and do not have systemic symptom onset will be included in covariate-adjusted analysis.

Determination of study drug blood level: Study drug levels will be measured via a liquid chromatography-tandem mass spectrometric (LC-MS/MS) assay method. The assay will be performed on a Shimadzu 8060 LC-MS/MS system, which is available at the Singapore General Hospital.

Gene expression studies: Gene expression in whole blood would be carried out using Nanostring nCounter assay. This assay provides a multiplex approach to identify the genes that the investigator have previously used to validate the hits from the microarray that identified adaptive ER stress as a susceptibility factor for symptomatic YF17D infection (see preliminary data). Importantly, the investigator have worked with Nanostring, to customize a comprehensive set of probes that are able to directly quantify mRNA transcripts in the ER stress and TCA cycle pathways, which would be the target genes in this trial. This approach is also chosen due to the CSA budget constraint. Nonetheless, the study team will collect extra clinical samples as backup and explore the use of RNAseq to discover the pharmacogenomics of metformin through additional funding from other grant sources.

This proposed gene expression study will be carried out at the Viral Research and Experimental Medicine Centre @ SingHealth Duke-NUS (ViREMiCS). ViREMiCS was established by the PI and collaborator, Eng Eong Ooi as a research centre in the SingHealth Duke-NUS Academic Medicine Centre partnership. It has established a suite of molecular and systems biology tools to support and accelerate proof-of concept clinical trials. The investigators thus do not anticipate any problem in using this approach to measure gene expression in blood samples.

Proteomics and Metabolomic profiling: Plasma metabolomics will be examined using capillary electrophoresis/mass spectrometry (CE/MS), and liquid chromatography/mass spectrometry LC-MS/MS as we have previously employed to measure the polar metabolites from glycolysis and TCA cycle [18, 25]. Proteomics will be measured using LC-MS/MS. These assays will be carried out using the core equipment available in the Programme in Emerging Infectious Diseases and Metabolomics Core Facility, both in Duke-NUS. This will enable a multi-omics approach to support enhanced biological insights.

Chemokine and Cytokine: Serum chemokine and cytokine levels will be measured using the Luminex or Olink assay that enables more than 40 serum chemokines and cytokines to be measured simultaneously.

YF Viremia and PRNT titres: YF viremia loads will be assessed using quantitative real-time PCR (qRT-PCR). Anti-YF neutralising antibody titres will be measured by plaque reduction neutralisation test (PRNT). Briefly, 50 PFU (plaque forming units) of YF17D virus will be incubated with 2-fold serial dilutions of human serum for one hour at 37oC, and then added to a monolayer of Vero cells in 24-well plates. One hour later, media will be aspirated and cells overlaid with carboxymethyl cellulose 1% in maintenance media. After 5 days, cells will be fixed, washed and stained with crystal violet. The number of plaques will be counted and PRNT50 titres determined using a sigmoid dose-response curve fit as reciprocal values.

scRNA-seq and T-cell Studies: Single cell RNA sequencing (scRNA-seq) will be performed on PBMCs isolated before and after metformin treatment to determine the impact of metformin treatment on different immune cell subsets. This proposed study will be carried out in collaboration with the Genome Biology Facility at Duke-NUS. Subsequently, using the findings of scRNA-seq as a guide, we will then assess T-cell function and activity using either flow cytometry or enzyme-linked immune absorbent spot (ELISPOT) assay. These assays will be carried out using core equipment available in the Programme in Emerging Infectious Diseases in Duke-NUS.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 21-40 years of age at time of screening
2. Body Mass Index of 20-25 kg/m2
3. No known drug allergies and are not currently receiving regular immune-modulating therapy such as metformin, NSAIDs, paracetamol, corticosteroids or statins.
4. Subjects who give written informed consent approved by the Ethical Review Board governing the site.
5. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
6. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening.
7. Negative for diabetes mellitus by HbA1c
8. Accessible vein at the forearm for blood collection.
9. Subjects who are willing to comply with the requirements of the study protocol and scheduled visits. (e.g., completion of the subject diary, return for follow-up visits) and who are willing to make themselves available for the duration of the study, with access to a consistent means of telephone contact, which may be either at home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e. a common-use phone serving multiple rooms or apartments).

Exclusion Criteria:

1. History of severe drug and/or food allergies and/or known allergies to the trial product or its components and any ingredients in the placebo pill.
2. Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.
3. Woman who is pregnant or breast feeding.
4. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders that would be a risk factor when administered the Investigational Product (IP).
5. Diagnosed with cancer or on treatment for cancer within the 3 years prior to the screening.
6. Evidence of clinically significant anemia and other any significant active hematological disease, or having donated > 450 mL of blood within the past three months.
7. Evidence of substance abuse, or previous substance abuse.
8. Participation in a study involving administration of an investigational compound within the past four months, or planned participation during the duration of this study.
9. Subjects who are on long term immune-modulating therapy (e.g. NSAIDs, Paracetamol, Corticosteroids, Statins etc.) for other medical condition for the last 6 months.
10. Subject who are on long term medication for concurrent medical conditions.
11. Administration of any licensed vaccine within 30 days before the first study vaccine dose.
12. Subject who has been vaccinated with YF vaccine previously.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic outcome | Day 0 to Day 18
  We will employ the definitions of systemic symptoms, based on the WHO guidelines for surveillance of YF vaccine-related AEs, and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 as previously published. For pain symptoms (i.e. headache, myalgia, arthralgia), a standardized Numerical pain Rating Scale (NRS) will be used. Subjects will be monitored over a 2-week period starting immediately after YF vaccination

SECONDARY OUTCOMES:
Reduction in pro-inflammatory and innate immune responses at day 1 post-infection | Day 0 to Day 32
  The rationale for this is that we have previously shown that expression of genes in these pathways at day 1 post-YF17D infection correlated with the development of symptoms at a median time of 6 days post-infection. Measurements of these genes will be done using the panel of Nanostring nCounter probes we have established in ViREMiCS.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny GH Low, MRCP (UK), Principal Investigator — Singapore General Hospital
Locations (1):
- Singhealth Investigational Medicine Unit, Singapore, Singapore

REFERENCES:
- [Background] Hueston L, Ramirez R, Mahalingam S. Enhancement of Zika Infection by Dengue Virus-Specific Antibody Is Associated With Low Levels of Antiviral Factors. J Infect Dis. 2017 Sep 1;216(5):612-614. doi: 10.1093/infdis/jix344. No abstract available. PMID 28931226
- [Background] Wang A, Luan HH, Medzhitov R. An evolutionary perspective on immunometabolism. Science. 2019 Jan 11;363(6423):eaar3932. doi: 10.1126/science.aar3932. PMID 30630899
- [Background] Lashley FR. Emerging infectious diseases at the beginning of the 21st century. Online J Issues Nurs. 2006 Jan 31;11(1):2. PMID 16629503
- [Background] Steinberg GR. Role of the AMP-activated protein kinase in regulating fatty acid metabolism during exercise. Appl Physiol Nutr Metab. 2009 Jun;34(3):315-22. doi: 10.1139/H09-009. PMID 19448692
- [Background] Jung TW, Choi KM. Pharmacological Modulators of Endoplasmic Reticulum Stress in Metabolic Diseases. Int J Mol Sci. 2016 Feb 1;17(2):192. doi: 10.3390/ijms17020192. PMID 26840310
- [Background] Cameron AR, Morrison VL, Levin D, Mohan M, Forteath C, Beall C, McNeilly AD, Balfour DJ, Savinko T, Wong AK, Viollet B, Sakamoto K, Fagerholm SC, Foretz M, Lang CC, Rena G. Anti-Inflammatory Effects of Metformin Irrespective of Diabetes Status. Circ Res. 2016 Aug 19;119(5):652-65. doi: 10.1161/CIRCRESAHA.116.308445. Epub 2016 Jul 14. PMID 27418629
- [Background] Vasamsetti SB, Karnewar S, Kanugula AK, Thatipalli AR, Kumar JM, Kotamraju S. Metformin inhibits monocyte-to-macrophage differentiation via AMPK-mediated inhibition of STAT3 activation: potential role in atherosclerosis. Diabetes. 2015 Jun;64(6):2028-41. doi: 10.2337/db14-1225. Epub 2014 Dec 31. PMID 25552600
- [Background] Badawi A, Velummailum R, Ryoo SG, Senthinathan A, Yaghoubi S, Vasileva D, Ostermeier E, Plishka M, Soosaipillai M, Arora P. Prevalence of chronic comorbidities in dengue fever and West Nile virus: A systematic review and meta-analysis. PLoS One. 2018 Jul 10;13(7):e0200200. doi: 10.1371/journal.pone.0200200. eCollection 2018. PMID 29990356
- [Background] Pichainarong N, Mongkalangoon N, Kalayanarooj S, Chaveepojnkamjorn W. Relationship between body size and severity of dengue hemorrhagic fever among children aged 0-14 years. Southeast Asian J Trop Med Public Health. 2006 Mar;37(2):283-8. PMID 17124987
- [Background] Karki S, Muscatello DJ, Banks E, MacIntyre CR, McIntyre P, Liu B. Association between body mass index and laboratory-confirmed influenza in middle aged and older adults: a prospective cohort study. Int J Obes (Lond). 2018 Aug;42(8):1480-1488. doi: 10.1038/s41366-018-0029-x. Epub 2018 Mar 7. PMID 29515210
- [Background] Bodmer M, Meier C, Krahenbuhl S, Jick SS, Meier CR. Metformin, sulfonylureas, or other antidiabetes drugs and the risk of lactic acidosis or hypoglycemia: a nested case-control analysis. Diabetes Care. 2008 Nov;31(11):2086-91. doi: 10.2337/dc08-1171. Epub 2008 Sep 9. PMID 18782901
- [Background] Preiss D, Lloyd SM, Ford I, McMurray JJ, Holman RR, Welsh P, Fisher M, Packard CJ, Sattar N. Metformin for non-diabetic patients with coronary heart disease (the CAMERA study): a randomised controlled trial. Lancet Diabetes Endocrinol. 2014 Feb;2(2):116-24. doi: 10.1016/S2213-8587(13)70152-9. Epub 2013 Nov 7. PMID 24622715
- [Background] Kaplowitz P. Is There a Role for Metformin in the Treatment of Childhood Obesity? Pediatrics. 2017 Jul;140(1):e20171205. doi: 10.1542/peds.2017-1205. Epub 2017 Jun 12. No abstract available. PMID 28759418
- [Background] Diabetes Prevention Program Research Group. Long-term safety, tolerability, and weight loss associated with metformin in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2012 Apr;35(4):731-7. doi: 10.2337/dc11-1299. PMID 22442396
- [Background] Monath TP, Cetron MS. Prevention of yellow fever in persons traveling to the tropics. Clin Infect Dis. 2002 May 15;34(10):1369-78. doi: 10.1086/340104. Epub 2002 Apr 25. PMID 11981733
- [Background] Monath TP, Nichols R, Archambault WT, Moore L, Marchesani R, Tian J, Shope RE, Thomas N, Schrader R, Furby D, Bedford P. Comparative safety and immunogenicity of two yellow fever 17D vaccines (ARILVAX and YF-VAX) in a phase III multicenter, double-blind clinical trial. Am J Trop Med Hyg. 2002 May;66(5):533-41. doi: 10.4269/ajtmh.2002.66.533. PMID 12201587
- [Background] Chan KR, Wang X, Saron WAA, Gan ES, Tan HC, Mok DZL, Zhang SL, Lee YH, Liang C, Wijaya L, Ghosh S, Cheung YB, Tannenbaum SR, Abraham SN, St John AL, Low JGH, Ooi EE. Cross-reactive antibodies enhance live attenuated virus infection for increased immunogenicity. Nat Microbiol. 2016 Sep 19;1(12):16164. doi: 10.1038/nmicrobiol.2016.164. PMID 27642668
- [Background] Kuleshov MV, Jones MR, Rouillard AD, Fernandez NF, Duan Q, Wang Z, Koplev S, Jenkins SL, Jagodnik KM, Lachmann A, McDermott MG, Monteiro CD, Gundersen GW, Ma'ayan A. Enrichr: a comprehensive gene set enrichment analysis web server 2016 update. Nucleic Acids Res. 2016 Jul 8;44(W1):W90-7. doi: 10.1093/nar/gkw377. Epub 2016 May 3. PMID 27141961
- [Background] Mahmoudabadi G, Milo R, Phillips R. Energetic cost of building a virus. Proc Natl Acad Sci U S A. 2017 May 30;114(22):E4324-E4333. doi: 10.1073/pnas.1701670114. Epub 2017 May 16. PMID 28512219
- [Background] Kaufman RJ, Malhotra JD. Calcium trafficking integrates endoplasmic reticulum function with mitochondrial bioenergetics. Biochim Biophys Acta. 2014 Oct;1843(10):2233-9. doi: 10.1016/j.bbamcr.2014.03.022. Epub 2014 Mar 30. PMID 24690484
- [Background] Wang M, Kaufman RJ. Protein misfolding in the endoplasmic reticulum as a conduit to human disease. Nature. 2016 Jan 21;529(7586):326-35. doi: 10.1038/nature17041. PMID 26791723
- [Background] Pryor WA, Jin X, Squadrito GL. One- and two-electron oxidations of methionine by peroxynitrite. Proc Natl Acad Sci U S A. 1994 Nov 8;91(23):11173-7. doi: 10.1073/pnas.91.23.11173. PMID 7972029
- [Background] Wang Y, Branicky R, Noe A, Hekimi S. Superoxide dismutases: Dual roles in controlling ROS damage and regulating ROS signaling. J Cell Biol. 2018 Jun 4;217(6):1915-1928. doi: 10.1083/jcb.201708007. Epub 2018 Apr 18. PMID 29669742
- [Background] Sung C, Wei Y, Watanabe S, Lee HS, Khoo YM, Fan L, Rathore AP, Chan KW, Choy MM, Kamaraj US, Sessions OM, Aw P, de Sessions PF, Lee B, Connolly JE, Hibberd ML, Vijaykrishna D, Wijaya L, Ooi EE, Low JG, Vasudevan SG. Extended Evaluation of Virological, Immunological and Pharmacokinetic Endpoints of CELADEN: A Randomized, Placebo-Controlled Trial of Celgosivir in Dengue Fever Patients. PLoS Negl Trop Dis. 2016 Aug 10;10(8):e0004851. doi: 10.1371/journal.pntd.0004851. eCollection 2016 Aug. PMID 27509020
- [Background] Cooper SA, Desjardins PJ, Turk DC, Dworkin RH, Katz NP, Kehlet H, Ballantyne JC, Burke LB, Carragee E, Cowan P, Croll S, Dionne RA, Farrar JT, Gilron I, Gordon DB, Iyengar S, Jay GW, Kalso EA, Kerns RD, McDermott MP, Raja SN, Rappaport BA, Rauschkolb C, Royal MA, Segerdahl M, Stauffer JW, Todd KH, Vanhove GF, Wallace MS, West C, White RE, Wu C. Research design considerations for single-dose analgesic clinical trials in acute pain: IMMPACT recommendations. Pain. 2016 Feb;157(2):288-301. doi: 10.1097/j.pain.0000000000000375. PMID 26683233
- [Background] Querec TD, Pulendran B. Understanding the role of innate immunity in the mechanism of action of the live attenuated Yellow Fever Vaccine 17D. Adv Exp Med Biol. 2007;590:43-53. doi: 10.1007/978-0-387-34814-8_3. No abstract available. PMID 17191376
- [Background] Ivashkiv LB, Donlin LT. Regulation of type I interferon responses. Nat Rev Immunol. 2014 Jan;14(1):36-49. doi: 10.1038/nri3581. PMID 24362405
- [Background] Yuan S, Chu H, Chan JF, Ye ZW, Wen L, Yan B, Lai PM, Tee KM, Huang J, Chen D, Li C, Zhao X, Yang D, Chiu MC, Yip C, Poon VK, Chan CC, Sze KH, Zhou J, Chan IH, Kok KH, To KK, Kao RY, Lau JY, Jin DY, Perlman S, Yuen KY. SREBP-dependent lipidomic reprogramming as a broad-spectrum antiviral target. Nat Commun. 2019 Jan 10;10(1):120. doi: 10.1038/s41467-018-08015-x. PMID 30631056
- [Background] Hapuarachchi HC, Koo C, Rajarethinam J, Chong CS, Lin C, Yap G, Liu L, Lai YL, Ooi PL, Cutter J, Ng LC. Epidemic resurgence of dengue fever in Singapore in 2013-2014: A virological and entomological perspective. BMC Infect Dis. 2016 Jun 17;16:300. doi: 10.1186/s12879-016-1606-z. PMID 27316694
- [Background] Guzman MG, Gubler DJ, Izquierdo A, Martinez E, Halstead SB. Dengue infection. Nat Rev Dis Primers. 2016 Aug 18;2:16055. doi: 10.1038/nrdp.2016.55. PMID 27534439
- [Background] Garcia G, Gonzalez N, Perez AB, Sierra B, Aguirre E, Rizo D, Izquierdo A, Sanchez L, Diaz D, Lezcay M, Pacheco B, Hirayama K, Guzman MG. Long-term persistence of clinical symptoms in dengue-infected persons and its association with immunological disorders. Int J Infect Dis. 2011 Jan;15(1):e38-43. doi: 10.1016/j.ijid.2010.09.008. Epub 2010 Nov 26. PMID 21112804
- [Background] Halsey ES, Williams M, Laguna-Torres VA, Vilcarromero S, Ocana V, Kochel TJ, Marks MA. Occurrence and correlates of symptom persistence following acute dengue fever in Peru. Am J Trop Med Hyg. 2014 Mar;90(3):449-56. doi: 10.4269/ajtmh.13-0544. Epub 2014 Jan 27. PMID 24470564
- [Background] Seet RC, Quek AM, Lim EC. Post-infectious fatigue syndrome in dengue infection. J Clin Virol. 2007 Jan;38(1):1-6. doi: 10.1016/j.jcv.2006.10.011. Epub 2006 Nov 29. PMID 17137834
- [Background] Teixeira Lde A, Lopes JS, Martins AG, Campos FA, Miranzi Sde S, Nascentes GA. [Persistence of dengue symptoms in patients in Uberaba, Minas Gerais State, Brazil]. Cad Saude Publica. 2010 Mar;26(3):624-30. doi: 10.1590/s0102-311x2010000300019. Portuguese. PMID 20464080
- [Background] Tristao-Sa R, Kubelka CF, Zandonade E, Zagne SM, Rocha Nde S, Zagne LO, Araujo NF, Amin B, Fazoli F, Souza LJ, Cruz OG, Cunha RV, Nascimento Dd, Froes IB, Nogueira RM. Clinical and hepatic evaluation in adult dengue patients: a prospective two-month cohort study. Rev Soc Bras Med Trop. 2012 Dec;45(6):675-81. doi: 10.1590/s0037-86822012000600004. PMID 23295867
- [Background] Tiga DC, Undurraga EA, Ramos-Castaneda J, Martinez-Vega RA, Tschampl CA, Shepard DS. Persistent Symptoms of Dengue: Estimates of the Incremental Disease and Economic Burden in Mexico. Am J Trop Med Hyg. 2016 May 4;94(5):1085-1089. doi: 10.4269/ajtmh.15-0896. Epub 2016 Mar 14. PMID 26976885